CLINICAL TRIAL: NCT03942562
Title: Temporal Relationship in Recovery of Muscular Pain, Functional Variables and Normal Gait Pattern in an Experimental Muscular Pain Model in Hamstrings
Brief Title: Temporal Relationship in Recovery of Muscular Pain and Functional Variables in an Experimental Muscular Pain Model in Hamstrings
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Other Study IDs: PI18/208
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Pain, Muscle
Keywords: DOMS; Healthy subjects; Pressure pain thresholds; Active Knee Extension test; Maximal strength; Electromyography; Plantar pressure measurement; Gait analysis
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Basal measurements are taken in relation to the study variables. Immediately subjects perform eccentric exercise on right hamstrings to develop delayed onset muscle soreness (DOMS).

Measurements of the study variables are taken in the same conditions 48, 96 and 168 hours after the exercise to study the evolution of the variables while recovering from DOMS.

DETAILED DESCRIPTION:
Basal measurements are taken in relation to the study variables.

The variables are:

* pressure pain thresholds
* electromyography values
* static and dynamic plantar pressure measurement
* active knee extensibility
* maximal strength of knee flexors
* thermography
* scales of pain perception

Immediately subjects perform eccentric exercise on right hamstrings to develop DOMS (delay onset muscle soreness).

Measurements of the study variables are taken in the same conditions 48, 96 and 168 hours after the exercise to study the evolution of the variables while recovering from DOMS.

ELIGIBILITY:
Inclusion Criteria:

* not sedentary subject (IPAQ scale > 600 MET)
* healthy subjects, without pain nor injury at the moment

Exclusion Criteria:

* subjects with acute or chronic pain on every spot of pelvis or lower limbs at the momento or for the last 3 months;
* subjects with history of severe injury in the hamstrings muscles;
* presence of serious illness;
* presence of pathologies in relation to chronic pain (as fibromyalgia, migraine disorders, non specific and chronic lumbar pain);
* not commitment for continuity in the study program;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Non sedentary healthy men
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in spatio temporal parameters of gait | Baseline, 48 hours, 96 hours, 1 week
  Changes in spatio temporal parameters of gait over a treadmill will be measurement using an optical measurement system consisting of a transmitting and receiving bar (OptoGait System).

SECONDARY OUTCOMES:
Changes in Pressure Pain Thresholds | Baseline, 48 hours, 96 hours, 1 week
  Changes in pressure pain thresholds (PPT) will be determined with pressure algometry bilaterally over the leg and shoulder. PPT is defined as the exact time point where the pressure is first being perceived at painful.
Changes in active knee extension test | Baseline, 48 hours, 96 hours, 1 week
  Changes in range of motion (°; degrees) will be assessed in both sides using the active knee extension (AKE) test.
  AKE test: subject is lying prone with hip and knee flexed at 90°. Then, maximal knee extension is performed.
Changes in knee-flexors maximal isometric muscle strength | Baseline, 48 hours, 96 hours, 1 week
  Changes in knee-flexors maximal isometric strength (Newton) will be assessed by using a hand-held dynamometer.
Electromyography (EMG) measurement during the tests | Baseline, 48 hours, 96 hours, 1 week
  Electromyography values will be taken from hamstrings during the performance of gait analysis and dynamometry
Changes in thermography on hamstrings areas | Baseline, 48 hours, 96 hours, 1 week
  A thermography image will be taken every day of assessment. Changes in colour pixels will be analysed to determine temperature changes.
Changes in static and dynamic plantar pressure measurement | Baseline, 48 hours, 96 hours, 1 week
  Changes in static and dynamic plantar pressure measurement will be performed in every session by using a pressure platform.
Changes in subjective perception of pain and impairment: Two questionnaire (Modified 7-item Likert Scales) | 48 hours, 96 hours, 1 week
  Two questionnaires (Modified 7-item Likert Scales) are filled up by the subject to show subjective perception of pain related to movement along the recovery period.
  Scale of pain intensity, from 0 (no pain) to 6 (higher pain intensity). Scale of functional impairment, from 0 (no impairment) to 6 (higher impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Víctor Doménech, MSc, Study Director — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
We don't plan to share data collected